CLINICAL TRIAL: NCT04249596
Title: Tianeptine for Treatment Resistant Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: Jonathan A. Javitch, MD, PhD (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Stanford University (Other)
Responsible Party: Sponsor-Investigator, Jonathan A. Javitch, MD, PhD, Professor of Psychiatry and of Pharmacology, New York State Psychiatric Institute
Organization: New York State Psychiatric Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7944/8436
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Treatment (Experimental): All subjects will be treated for 8 weeks of treatment with Tianeptine (Tianeurax 12.5 mg) 3 times a day (9am, 1pm, 5pm).
  Interventions: Drug: Tianeptine Sodium

INTERVENTIONS:
Drug: Tianeptine Sodium — At baseline, and following 8 weeks of treatment with tianeptine(12.5 mg, 3x daily), participants will be assessed in a number of procedures to evaluate their emotional and physical pain state and pain stimulus response and the relationship of such states/responses to endogenous opioid signaling. To further assess emotional pain, participants will also undergo fMRI while performing a validated social rejection and social acceptance paradigm known to induce endogenous opioid release in control subjects and blunted release in MDD. Examining both rejection and acceptance is important because the MOR system regulates both social distress and social reward in animals and humans, and tianeptine may also act on abnormal MOR-mediated responses to social acceptance in MDD. Likewise, a second fMRI scan will be used to explore physical pain response using an established thermal pain sensitivity task. The protocol at Stanford University will not include pain testing or imaging studies.
  Other Names: Tianeurex 12.5 mg

SUMMARY:
The studies will be conducted in parallel at two sites: the the Mood and Anxiety Disorders Program at the Icahn School of Medicine at Mount Sinai (MSSM), and Stanford Depression Research Clinic at Stanford University School of Medicine (SUSM). In addition, MRI studies for the MSSM patients will be carried out at the New York State Psychaitric Institute (NYSPI). The following procedures will be approved by the local Institutional Review Boards (IRBs) at each site, where the site PIs (Alla Landa, PhD, NYSPI, James Murrough, MD at MSSM, and Alan Schatzberg, MD at SUSM) will be responsible for overseeing conduct of the study at their respective site. Dr. Jonathan Javitch is the scientific leader of this program and holds the IND for tianeptine use in this study.

Investigators will recruit 75 participants with current unipolar MDD, non-delusional, between 21-60, who have failed at least 2 two adequate treatment trials with a standard antidepressant. Patients will receive an 8-week treatment trial of tianeptine. MSSM patients will also undergo structural and task-based magnetic resonance imaging (MRI) that will be performed under Dr. Landa's direction at NYSPI in order to maintain the internal validity of the data set. MSSM subjects will be transported to NYSPI to complete neuroimaging procedures as described below. Participants will be screened for MRI clearance during their screening visit and again at NYSPI on the day of the scan. Subjects will be asked MRI screening questions to ensure that are scanning eligible. Participants will also have additional tubes of blood drawn for human whole-genomic testing. This microarray will be used to identify regions of the human genome that contribute to disease susceptibility and phenotypes. The Illumina human whole-genome array will be used to provide a comprehensive view of the genome, detects single nucleotide polymorphisms and other variations across the genome.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a leading cause of disability in adults worldwide (~16M patients in United States alone). Unfortunately, only 35-40% of patients achieve full remission following first-line treatment and treatment-resistant depression (TRD), failure to respond to 2 or more treatments, is a critical clinical problem. As with MDD, there is mechanistic heterogeneity in TRD and consequently, there is a need to develop treatments targeted to biologically distinct subgroups of patients. Significant evidence suggests dysfunction of endogenous opioid signaling pathways as a key biological deficit in some MDD patients. Investigators hypothesize that a subgroup of MDD patients with deficient opioid receptor signaling who have failed previous trials of antidepressants will better respond to pharmacological interventions specifically targeting this biological mechanism.

In this application, Investigators propose to target the mu-opioid receptor (MOR) in TRD patients by using the antidepressant tianeptine. Although not available in the United States, Tianeptine is an atypical antidepressant that has been used clinically in Europe, Asia, and South America since the late 1980s in millions of patients. Until recently tianeptine's molecular mechanism of action had remained unknown. Tianeptine is a different type of antidepressant than those currently approved in the United States in that it has a different mechanism of action than other antidepressants. Tianeptine is an opioid antagonist; it binds at the mu-opioid receptor. Currently approved antidepressants act on other systems of the brain that primarily affect serotonin, norepinephrine, and dopamine. Work in our laboratories has shown that tianeptine acts as a selective agonist of MOR, signaling in a manner analogous to enkephalins and endorphins, the endogenous opioid peptides. The investigator applied for and received an IND to import and use tianeptine for this study.

The studies will be conducted in parallel at two sites: the the Mood and Anxiety Disorders Program at the Icahn School of Medicine at Mount Sinai (MSSM), and Stanford Depression Research Clinic at Stanford University School of Medicine (SUSM). In addition, MRI studies for the MSSM patients will be carried out at the New York State Psychaitric Institute (NYSPI). The following procedures will be approved by the local Institutional Review Boards (IRBs) at each site, where the site PIs (Alla Landa, PhD, NYSPI, James Murrough, MD at MSSM, and Alan Schatzberg, MD at SUSM) will be responsible for overseeing conduct of the study at their respective site. Dr. Jonathan Javitch is the scientific leader of this program and holds the IND for tianeptine use in this study.

Investigators will recruit 75 participants with current unipolar MDD, non-delusional, between 21-60, who have failed at least 2 two adequate treatment trials with a standard antidepressant. MSSM patients will also undergo structural and task-based magnetic resonance imaging (MRI) that will be performed under Dr. Alla Landa's direction at NYSPI in order to maintain the internal validity of the data set. MSSM subjects will be transported to NYSPI to complete neuroimaging procedures as described below. Participants will be screened for MRI clearance during their screening visit and again at NYSPI on the day of the scan. Subjects will be asked MRI screening questions to ensure that are scanning eligible. Participants will also have additional tubes of blood drawn for human whole-genomic testing. This microarray will be used to identify regions of the human genome that contribute to disease susceptibility and phenotypes. The Illumina human whole-genome array will be used to provide a comprehensive view of the genome, detects single nucleotide polymorphisms and other variations across the genome.

The major goals of this project are (1) to determine if tianeptine is an effective antidepressant in patients who have failed two previous trials, (2) to define the relationship between opioid signaling deficits and response to tianeptine treatment, and (3) to develop a comprehensive assessment battery capable of identifying endogenous opioid signaling deficits to explore biological heterogeneity in the TRD population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 - 60 years, male or female
2. Current diagnosis of Major Depressive Disorder (MDD) without psychotic features
3. 24-item Hamilton Rating Scale for Depression (HRSD) ≥ 16
4. At least two previous antidepressant treatment failures (adequate trials within current episode) with a SSRI, SNRI, bupropion, tricyclic antidepressant, mirtazapine, nefazodone, or monoamine oxidase inhibitor, or transcranial magnetic stimulation (TMS), or IV ketamine or nasal ketamine.
5. Capable of providing informed consent and complying with study procedures
6. Currently using or willing to use contraception, if woman of childbearing potential (such as condoms, IUD, or oral contraceptive), for duration of the study.

Exclusion Criteria:

1. Any history of opioid-use disorder
2. Any history of moderate- non-opioid (except for Nicotine) substance-use disorder.
3. Any severity of alcohol use disorder (including mild)
4. Past or current psychosis, psychotic disorder (including psychotic MDD), mania, or bipolar disorder
5. Hamilton Rating Scale for Depression (HRSD) suicide item > 2 or Clinical Global Impressions (CGI)-Severity score of 7 at baseline
6. Previous or current treatment with Tianeptine
7. Current treatment or currently taking an opioid.
8. Failed depression treatment with electroconvulsive therapy.
9. Acute, severe, or unstable medical illness
10. Weight > 300 lbs, or girth size incompatible with scanner bore.
11. Any physical or intellectual disability adversely affecting ability to complete assessments. MMSE <26
12. for MSSM site - Having contraindication to MRI scanning (such as metal in body) or inability to tolerate the scanning procedures (e.g., severe obesity, claustrophobia)
13. Current pregnancy or currently breast feeding.
14. Abnormal baseline liver function tests
15. Currently being treated with an antidepressant medication, an antipsychotic or mood stabilizer.

    a) If a participant is taking a protocol dis-allowed medication at the time of screening and despite medication treatment still meets the inclusion criteria of an HRSD>16, the participant may discontinue the medication under the supervision of their treating physician or the study clinician.
16. Positive urine toxicity at screening (except for cannabinoid)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alla Landa, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (3):
- United States (3):
  - Stanford Depression Research Clinic at Stanford University School of Medicine, Stanford, California
  - Mood and Anxiety Disorders Program at the Icahn School of Medicine at Mount Sinai, New York, New York
  - New York State Psychiatric Institute, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from outpatient clinics at three academic medical centers: New York State Psychiatric Institute, Icahn School of Medicine at Mount Sinai, and Stanford University. Recruitment occurred from October 2020 to August 2024. Study was terminated early due to inadequate recruitment (38 of 75 target enrolled).
Pre-assignment Details: Baseline assessments (HAMD-24, ARSQ) were performed prior to treatment initiation. Participants on antidepressants completed a taper period before baseline. Some participants who consented did not initiate treatment due to screen failure, consent withdrawal, or loss to follow-up during the screening period. Per protocol, enrollment was defined as initiation of study medication; participants who did not receive study drug were not considered enrolled.
Groups:
- Tianeptine Sodium 12.5mg TID Treatment: Open-label tianeptine sodium 12.5mg three times daily for 8 weeks
Period: Overall Study
Arm/Group | Tianeptine Sodium 12.5mg TID Treatment
Started | 38
Completed | 30
Not Completed | 8
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study medication
Arm/Group | Tianeptine Sodium 12.5mg TID Treatment
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.2 (10.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 23
  Male | 14
  Non-binary | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 4
  Unknown or Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 4
  Unknown or Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 2
Baseline HAMD-24 Score [Mean (Standard Deviation); unit: units on a scale] — Hamilton Rating Scale for Depression, 24-item. Range 0-74, higher scores indicate greater severity.
  units on a scale | 25.4 (5.8)
Baseline ARSQ Score [Mean (Standard Deviation); unit: units on a scale] — Adult Rejection Sensitivity Questionnaire (A-RSQ; Berenson et al., 2009). Measures rejection sensitivity, the disposition to anxiously expect, readily perceive, and intensely react to rejection. Respondents rate 9 situations on rejection concern (1-6) and acceptance expectancy (1-6). Item scores = rejection concern × (7 - acceptance expectancy). Total score is the mean of 9 item scores. Range: 1-36; higher scores indicate greater rejection sensitivity.
  units on a scale | 14.6 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression, 24-item (HAMD-24)
Description: Our target is depressive symptomatology as measured by the Hamilton Rating Scale for Depression (HRSD). The HRSD is a 24-item questionnaire used as an indication of depression and a guide to evaluate recovery. Total scores range from 0-74, not including atypical symptoms sub-scale. A score of 16 or above is typically considered to indicate the presence of depressive symptoms. Higher scores indicate greater severity.
Time Frame: 8 weeks
Population: Participants who completed 8-week treatment protocol (30 of 38 who started)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tianeptine Sodium 12.5mg TID Treatment
Number analyzed (Participants) | 30
units on a scale | -5.2 (9.8)

2. Secondary Outcome: Response Rate
Description: Proportion of participants achieving ≥50% reduction in HAMD-24 score from baseline
Time Frame: 8 weeks
Population: Participants who completed 8-week treatment protocol (30 of 38 who started)
Measure: Count of Participants; unit: Participants
Arm/Group | Tianeptine Sodium 12.5mg TID Treatment
Number analyzed (Participants) | 30
Participants | 7

3. Secondary Outcome: Remission Rate
Description: Proportion of participants achieving HAMD-24 score ≤10 at Week 8
Time Frame: 8 weeks
Population: Participants who completed 8-week treatment protocol (30 of 38 who started)
Measure: Count of Participants; unit: Participants
Arm/Group | Tianeptine Sodium 12.5mg TID Treatment
Number analyzed (Participants) | 30
Participants | 6

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse events were assessed at each study visit using systematic inquiry
Arm/Group | Tianeptine Sodium 12.5mg TID Treatment
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 1/38
Other Adverse Events (participants affected / at risk) | 4/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tianeptine Sodium 12.5mg TID Treatment (N=38)
Depression worsening requiring hospitalization (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tianeptine Sodium 12.5mg TID Treatment (N=38)
Headache (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 3

LIMITATIONS AND CAVEATS:
Study terminated early due to inadequate recruitment (38 of 75 target enrollment). Open-label, single-arm design without placebo control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT04249596/Prot_SAP_000.pdf